CLINICAL TRIAL: NCT04429191
Title: A Phase 1a/b Study to Evaluate the Safety & Tolerability of JSP191 in Combination With a Regimen of Low Dose Radiation & Fludarabine in Subjects With MDS or AML Undergoing Hematopoietic Cell Transplantation (HCT)
Brief Title: JSP191 Antibody Conditioning Regimen in MDS/AML Subjects Undergoing Allogenic Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jasper Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSP-CP-003
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: MYELODYSPLASTIC SYNDROME; MDS; ACUTE MYELOID LEUKEMIA; AML
Keywords: ACUTE MYELOID LEUKEMIA; AML; MDS; MYELODYSPLASTIC SYNDROME
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blood Stem Cell Transplant w/ anti-CD117 conditioning (Experimental): The phase 1a portion of the study plans to assess approximately 3 planned dose cohorts of JSP191: 0.3 mg/kg, 0.6 mg/kg, and 1.0 mg/kg to determine the maximum tolerated dose for expansion. Subjects will receive a single dose of intravenous JSP191 antibody followed by monitoring for antibody clearance. Once the antibody has cleared below a certain level, patients will receive stem cell transplant and be monitored for hematopoietic recovery.
  The phase 1b portion of the study will enroll additional subjects at the expansion dose in order to further explore the safety, feasibility, and PK of that dose.
  Interventions: Biological: Humanized anti-CD117 Monoclonal Antibody (JSP191)

INTERVENTIONS:
Biological: Humanized anti-CD117 Monoclonal Antibody (JSP191) — Procedure: single intravenous infusion of JSP191 antibody
  Other Names: JSP191

SUMMARY:
This is a Phase 1a/b study to evaluate the safety and tolerability of an antibody conditioning regimen known as JSP191, in combination with low dose radiation and fludarabine, in subjects with Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML) undergoing allogenic blood stem cell transplantation.

DETAILED DESCRIPTION:
This is a Phase 1a/b study to evaluate the safety and tolerability of an antibody conditioning regimen known as JSP191, in combination with low dose radiation and fludarabine in subjects with Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML) undergoing allogenic blood stem cell transplantation.

Blood Stem Cell transplantation offers the only potentially curative therapy for many forms of Acute Myeloid Leukemia (AML) and for Myelodysplastic Syndrome (MDS). While standard of care conditioning regimens given prior to blood Stem Cell transplantation, such as standard TBI/Flu conditioning are well tolerated, they are associated with increased rates of relapse due to persistence of disease causing Hematopoietic Stem Cells and insufficient graft versus leukemia effect.

The biological conditioning regimen JSP191 is an antibody that binds to CD117. CD117 is the receptor for Stem Cell Factor on blood forming cells. CD117 binding to Stem Cell Factor is critical for survival and maintenance of blood forming stem cells.

The binding of JSP191 to CD117 blocks CD117 from binding to Stem Cell Factor on blood forming stem cells. In the absence of CD117/Stem Cell Factor binding, hematopoietic stem cells that are currently occupying the bone marrow niches in MDS/AML patients are depleted.

This study will investigate the safety and tolerability of adding JSP191 (an anti-CD117 monoclonal antibody therapy) to standard TBI/Flu conditioning regimen in adults with AML and MDS undergoing hematopoietic stem cell transplant.

ELIGIBILITY:
Key Inclusion Criteria:

* AML/MDS as defined by specific criteria, including but not limited to the following subtypes:

  1. AML in CR
  2. MDS < 5% BM blasts
  3. MDS 5 - 10% BM blasts
  4. AML not in CR or MDS > 10% BM blasts
* Patients with human leukocyte antigen (HLA) matched related or unrelated donors
* Adequate end organ function as defined in study protocol

Key Exclusion Criteria:

* Patients with any acute or uncontrolled infections
* Patients receiving any other investigational agents
* Patients with active non-hematologic malignancy
* Prior allogeneic hematologic cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-12-08 (Estimated)

PRIMARY OUTCOMES:
The number of subjects experiencing adverse events and serious adverse events will be assessed. | Up to 1 year post Donor Cell Transplant (28 days dose limiting toxicity period)
  The number of subjects experiencing adverse events and serious adverse events will be assessed.
The number of dose limiting toxicities will be assessed. | Up to 1 year post Donor Cell Transplant (28 days dose limiting toxicity period)
  The number of dose limiting toxicities will be assessed.
The type of dose limiting toxicities will be assessed. | Up to 1 year post Donor Cell Transplant (28 days dose limiting toxicity period)
  The type of dose limiting toxicities will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Muffly, MD,MS, Principal Investigator — Stanford University; Andrew Artz, MD,MS, Principal Investigator — City of Hope Medical Center; Bart Scott, MD, Principal Investigator — Fred Hutchinson Cancer Center; Catherine Lee, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah; Arpita Gandhi, MD, Principal Investigator — Oregon Health and Science University; Ankur Varma, MD,PhD, Principal Investigator — Rush University Medical Center
Locations (6):
- United States (6):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Stanford University, Stanford, California
  - Rush University Medical Center, Chicago, Illinois
  - Oregon Health & Science University, Portland, Oregon
  - Huntsman Cancer Institute - University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No